CLINICAL TRIAL: NCT01418248
Title: Evaluation of Exercise Intolerance and Right Heart Function in Patients With Heart Failure and Pulmonary Vascular Disease
Brief Title: Study of Exercise and Heart Function in Patients With Heart Failure and Pulmonary Vascular Disease
Acronym: EXEC
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Barry Borlaug, MD, Mayo Clinic
Other Study IDs: 11-004186
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Exercise Tolerance; Dyspnea; Heart Failure; Pulmonary Hypertension
Keywords: cardiac catheterization; echocardiography
MeSH Terms: conditions — Dyspnea; Heart Failure; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Heart Failure with Preserved Ejection Fraction (HFpEF) and Pulmonary Hypertension (PH) can be diagnosed noninvasively by Exercise Echocardiography (ExE) and Cardiopulmonary Exercise Testing (CPX) as compared with gold standard invasive hemodynamic assessment.

DETAILED DESCRIPTION:
* The broad objective of this proposal is to characterize the dynamic changes in cardiopulmonary mechanics during stress in patients with exertional dyspnea, establishing a comprehensive multimodality diagnostic approach to the evaluation of exercise intolerance.
* The specific objective is to prospectively compare established and novel parameters derived from echocardiography and CPX with simultaneous, gold standard invasive measures of cardiovascular hemodynamics at rest and with exercise stress to define the role of noninvasive testing in the diagnostic workup.
* The primary hypothesis is that combined ExE and CPX can noninvasively identify HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* exertional intolerance/dyspnea of unknown etiology
* referral to cardiac catheterization laboratory
* undergoing invasive hemodynamic evaluation for clinical purposes

Exclusion Criteria:

* hypertrophic cardiomyopathy
* constrictive pericarditis
* infiltrative myopathy (e.g. amyloid)
* congenital heart disease
* resting LVEF <50%
* > moderate mitral annular calcification
* moderate or greater left-sided valvular stenosis or regurgitation
* prior valve surgery
* basal septal wall motion abnormalities
* >70% epicardial coronary artery stenosis
* right ventricular infarction
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac Catheterization Laboratory
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic Utility ExE and CPX | Same day as clinically indicated Right Heart Catheterization (RHCath)

SECONDARY OUTCOMES:
Multiple integrated measures of cardiovascular function derived from RHCath, ExE and CPX along with rest/exercise natriuretic peptide levels | Same day as clinically indicated RHCath

CONTACTS AND LOCATIONS:
Overall Officials: Barry Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Obokata M, Kane GC, Sorimachi H, Reddy YNV, Olson TP, Egbe AC, Melenovsky V, Borlaug BA. Noninvasive evaluation of pulmonary artery pressure during exercise: the importance of right atrial hypertension. Eur Respir J. 2020 Feb 12;55(2):1901617. doi: 10.1183/13993003.01617-2019. Print 2020 Feb. PMID 31771997
- [Derived] Obokata M, Kane GC, Reddy YNV, Melenovsky V, Olson TP, Jarolim P, Borlaug BA. The neurohormonal basis of pulmonary hypertension in heart failure with preserved ejection fraction. Eur Heart J. 2019 Dec 1;40(45):3707-3717. doi: 10.1093/eurheartj/ehz626. PMID 31513270
- [Derived] Obokata M, Reddy YNV, Melenovsky V, Kane GC, Olson TP, Jarolim P, Borlaug BA. Myocardial Injury and Cardiac Reserve in Patients With Heart Failure and Preserved Ejection Fraction. J Am Coll Cardiol. 2018 Jul 3;72(1):29-40. doi: 10.1016/j.jacc.2018.04.039. PMID 29957229
- [Derived] Obokata M, Kane GC, Reddy YN, Olson TP, Melenovsky V, Borlaug BA. Role of Diastolic Stress Testing in the Evaluation for Heart Failure With Preserved Ejection Fraction: A Simultaneous Invasive-Echocardiographic Study. Circulation. 2017 Feb 28;135(9):825-838. doi: 10.1161/CIRCULATIONAHA.116.024822. Epub 2016 Dec 30. PMID 28039229
- [Derived] Andersen MJ, Hwang SJ, Kane GC, Melenovsky V, Olson TP, Fetterly K, Borlaug BA. Enhanced pulmonary vasodilator reserve and abnormal right ventricular: pulmonary artery coupling in heart failure with preserved ejection fraction. Circ Heart Fail. 2015 May;8(3):542-50. doi: 10.1161/CIRCHEARTFAILURE.114.002114. Epub 2015 Apr 9. PMID 25857307
- [Derived] Kobashigawa J, Patel J, Azarbal B, Kittleson M, Chang D, Czer L, Daun T, Luu M, Trento A, Cheng R, Esmailian F. Randomized pilot trial of gene expression profiling versus heart biopsy in the first year after heart transplant: early invasive monitoring attenuation through gene expression trial. Circ Heart Fail. 2015 May;8(3):557-64. doi: 10.1161/CIRCHEARTFAILURE.114.001658. Epub 2015 Feb 19. PMID 25697852
- [Derived] Andersen MJ, Olson TP, Melenovsky V, Kane GC, Borlaug BA. Differential hemodynamic effects of exercise and volume expansion in people with and without heart failure. Circ Heart Fail. 2015 Jan;8(1):41-8. doi: 10.1161/CIRCHEARTFAILURE.114.001731. Epub 2014 Oct 23. PMID 25342738